CLINICAL TRIAL: NCT05473143
Title: Proactive Prescription-based Fluid Management vs Usual Care in Critically Ill Patients on Kidney Replacement Therapy
Acronym: Probe-Fluid
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-02-2023-10829
Record Dates: First submitted 2022-07-15; First posted 2022-07-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Kidney Replacement; Critical Illness
Keywords: Fluid balance management; Ultrafiltration
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protocolized fluid removal (Experimental)
  Interventions: Other: Protocol-based fluid management
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Protocol-based fluid management — Fluid removal will be prescribed using a standardized template updated at least once per working day, before noon of each day, by the attending care team. This protocolized prescription will contain three components. Fluid removal will be prescribed using a standardized template updated at least once per working day, before noon of each day, by the attending care team. This protocolized prescription will contain three components.
  The first component of this prescription will be to define the 24h-fluid balance target either aiming for a negative fluid balance of 2 to 3% body weight (1.4-2.1 liters in a 70 Kg participant) (Option 1) or by aiming to avoid fluid accumulation by targeting a neutral fluid balance within 0.5% of body weight variation (-350 to +350 mL in a 70 Kg participant) (Option 2).
  The second component is to pre-specify a prescription for fluid removal using KRT.
  The third component is to prompt a daily re-evaluation of fluid intake by the attending care team.
  Arms: Protocolized fluid removal
Other: Usual care — The net fluid removal and the rate of net fluid removal will not be protocolized and will be prescribed and adjusted according to the attending care team without any specific guidance. The use of the documents provided for the intervention group will not be permitted in the control arm.
  Arms: Usual care

SUMMARY:
A pilot randomized clinical trial comparing a protocol-based fluid management strategy to usual care in critically ill patients receiving kidney replacement therapy. The fluid management protocol is intended to achieve neutral or negative daily fluid balance by both preventing and treating fluid accumulation.

DETAILED DESCRIPTION:
Severe acute kidney injury (AKI) in the intensive care unit (ICU) is almost uniformly complicated by fluid accumulation, thus making fluid removal a central component of the renal replacement therapy (KRT) prescription. Whereas the achievement and maintenance of euvolemia are critical objectives in the care of critically ill patients with severe AKI, there remain important knowledge gaps in our ability to effectively and safely deliver ultrafiltration. Multisystemic congestion resulting from fluid accumulation is believed to mediate adverse outcomes in this population and the timely use of mechanical fluid removal may improve prognosis. However, fluid removal may be associated with hemodynamic instability during KRT which may precipitate complications. The optimal fluid management strategy is currently unknown.

The study is a pilot randomized clinical trial comparing a protocol-based fluid management strategy with usual care in critically ill patients receiving KRT. The fluid management protocol is intended to achieve neutral or negative daily fluid balance by both preventing and treating fluid accumulation. The protocol was designed to provide a standardized framework to prescribe fluid removal while allowing the attending care team to modify treatment targets according to their clinical evaluation.

The primary objective of this trial is to determine whether the intervention results in a difference in cumulative fluid balance from randomization to 5 days. Feasibility will be documented including the ability to enroll the target population, protocol adherence, and the capacity to achieve follow-up through 90 days. Secondary outcomes will also include short-term patient outcomes, safety outcomes, and health resource utilization related to KRT delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admitted to the ICU
3. AKI during current hospitalization defined by the Kidney Disease: Improving Global Outcomes (KDIGO) criteria(1) as any of the following: Increase in serum creatinine by 27 µmol/L or more within any 48-hour window, or an increase in serum creatinine to 1.5 times baseline or more within the last 7 days, or a urine output less than 0.5 mL/kg/h for 6 hours.
4. Planned initiation of KRT within the following 12 hours or the receipt of KRT for AKI for ≤48 hours

Exclusion Criteria:

1. Lack of commitment to maintain kidney, pharmacologic or respiratory support at the time of screening, or probable transition to comfort care within 48 hours according to the treating physician
2. Probable discharge from the ICU within the next 48 hours according to treating physician
3. Severe burn injury (>10% of body surface area)
4. Severe abnormality in serum sodium (>155 or <120 mmol/L)
5. Important ongoing fluid losses are present and/or are expected to require continued maintenance IV fluids uring the next 48 hours
6. The clinical care team believes that the proposed intervention is inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative fluid balance | From randomization to the end of day 5
  The difference between quantifiable fluid intake and output

SECONDARY OUTCOMES:
Feasibility: Ability to successfully enroll | During screening and enrolment
  Target >30% of fully eligible patients
Feasibility: Protocol adherence | From randomization to the end of day 5
  defined as >80% of participants adhering to the allocated treatment for 5 days after enrolment
Feasibility: Ability to achieve follow-up | From randomization through day 90.
  Ability to achieve > 95% follow-up regarding all clinical outcomes
Clinical: Death | From randomization through day 90.
  Death from any cause
Clinical: Vasoactive therapy-free days | From randomization through day 28.
  A vasoactive-free day will be defined as ≥ 2 hours of receipt of any vasoactive therapy provided by continuous infusion within a 24 hour period. Vasoactive therapy include norepinephrine, vasopressin, phenylephrine, epinephrine, dopamine >5mcg/kg/min, and angiotensin II.
Clinical: Mechanical ventilation-free days | From randomization through day 28.
  A ventilator-free day will be defined as the receipt of ≥ 2 hours of mechanical ventilation within a 24-hour period.
Clinical: KRT-free days | From randomization through day 28.
  An KRT-free day will be defined receiving any KRT modality for ≥ 2 hours within a 24 hours period.
Clinical: ICU-free days | From randomization through day 90
  An ICU-free day will be defined as admission to an ICU for ≥ 2 hours within a 24 hours period.
Clinical: Hospital-free days | From randomization through day 90
  Hospital-free days will be defined as a 24-hour period completely free of an inpatient hospitalization.
Dependence on KRT | within +/- 7 days of the 90-day time point following randomization.
  KRT dependence will be defined by the receipt of any form of KRT
Resource use: cumulative time of continuous KRT | From randomization to the end of day 5
  Total cumulative duration in hours
Resource use: cumulative time of intermittent KRT | From randomization to the end of day 5
  Total cumulative duration in hours
Safety: Maximal vasopressor requirements | From randomization to the end of day 5
  Maximal vasopressor requirements as per the vasoactive-inotropic score recorded during each 24-hour period.
Safety: Severity of illness | From randomization to the end of day 5
  Total sequential organ failure assessment (SOFA) score recorded during each 24-hour period.
Process measures: Target fluid balance as prescribed in the initial fluid balance prescription for the day | From randomization to the end of day 5
Process measures: Proportion of time in which a neutral fluid balance target is selected by the clinical care team | From randomization to the end of day 5
Process measures: Clinical elements used to assess fluid accumulation | From randomization to the end of day 5
Process measures: The difference between the original target and the fluid balance achieved at the end of each 24-hour period | From randomization to the end of day 5

CONTACTS AND LOCATIONS:
Overall Officials: William Beaubien-Souligny, MD PhD, Study Chair — CHUM; Ron Wald, MDCM MPH, Study Chair — Unity Health Toronto; Sean Bagshaw, MD MSc, Study Chair — University of Alberta
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen A, Bouchard J, Neyra JA, Lamontagne F, Cote JM, Clark EG, da Costa BR, Gallagher M, Adhikari NKJ, Silver SA, Suri RS, Ostermann M, Neto AS, Bellomo R, Bagshaw SM, Wald R, Beaubien-Souligny W. Proactive Prescription-Based Fluid Management Versus Usual Care in Critically Ill Patients on Kidney Replacement Therapy (Probe-Fluid): A Pilot Clinical Trial Protocol. Can J Kidney Health Dis. 2025 Dec 9;12:20543581251391877. doi: 10.1177/20543581251391877. eCollection 2025. PMID 41393271